CLINICAL TRIAL: NCT00815776
Title: Treatment Outcome of Temporomandibular Disorders Via the Clayton Intra-aural Device (CID): A Randomized Clinical Trial
Brief Title: Treatment Outcomes for Temporomandibular Disorders (TMD) Via the Clayton Intra-aural Device (CID) Clinical Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ascentia Health, Inc. (Industry)
Responsible Party: Lawrence G. Clayton, Ascentia Health, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CID2007
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Results first posted 2010-08-06 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Temporomandibular Disorders
Keywords: Temporomandibular disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Treatment group receiving the CID
  Interventions: Device: Clayton Intra-aural Device (CID)
- 2 (Active Comparator): Group assigned a mouth splint
  Interventions: Device: Mouth Splint
- Exercise Control Group (Active Comparator): Group who received no device but were instead assigned a study-specified jaw exercise program
  Interventions: Other: Exercise Group

INTERVENTIONS:
Device: Clayton Intra-aural Device (CID) — The CID is a patented small, hollow, ear insert made of medical grade polymers that is custom-fit to each subject's ear. Each subject that is randomized to the CID study group will wear a pair of inserts, one in each ear. (For the purpose of this protocol, the pair of inserts will be referred to as the "CID").
  Arms: 1
Device: Mouth Splint — Group 2 subjects will be assigned to the active control device, which is current standard of care therapy. The device is an intraoral flat-planed splint full coverage plastic (hard) orthotic that fits over the occlusal one-third surfaces of the dentition. The appliance is made by taking a standard wax bite registration and is made using the standard technique of taking alginate impressions of the subject's teeth, pouring dental laboratory stone into the impression and processing the acrylic appliance on the stone model. This appliance raises the plane of occlusion and provides complete contact with the opposing dentition.
  Arms: 2
Other: Exercise Group — Subjects assigned to Group 3 will be asked to track daily compliance with the protocol-specific exercise plan in their 4 week diaries. The exercise plan will consist of the following instructions: subjects will be instructed to open their jaw as far as possible, without pain and hold the jaw in that position for 5 seconds. Subjects will then close their jaw and rest 10 seconds. The exercise should be repeated exactly ten times in a row, with a 10 second rest in between each stretch. Subjects will be advised to apply a warm compress to the jaw area after completing their exercises for 10 minutes.
  Arms: Exercise Control Group

SUMMARY:
The purpose of this study is to characterize the safety profile and assess the effectiveness of the CID in treating subjects with temporomandibular disorders (TMDs). This study is an open-label, three arm, randomized, unblinded clinical trial with a pre-treatment screening phase, a baseline visit and a 3 month treatment or exercise phase.

DETAILED DESCRIPTION:
After providing consent, subjects will be assessed as to whether they meet inclusion criteria for the study. Subjects will complete a 4 week diary to measure TMD symptoms by recording pain levels on a Visual Analog Scale (VAS) twice daily. Standardized Research Diagnostic Criteria (RDC) are used to classify types of TMDs. The formal assessment tool is known as the RDC/TMD. It is an empirically-based and operationalized system for diagnosing and classifying RDC/TMD using a biopsychosocial model of disease as a framework. The CMI/TMD(hereafter referred to as the CMI) is designed to provide a basis for evaluating the severity of TMD signs and symptoms. The CMI score is calculated from a dysfunction index (DI) and palpation index (PI). The majority of questions found in the CMI are also included in the RDC/TMD, with the exception of five questions. As part of the baseline medical history, all subjects will be asked the five questions that are included in the RDC/TMD but not included in the CMI. Data from the CMI and the five RDC/TMD questions will be combined in the database and scored according to scoring guidelines for the RDC/TMD in order to diagnose and classify TMDs for all study subjects. Subjects may be categorized in one or more of the three diagnostic groups, including muscle disorders (myofascial pain), arthralgia, and disc displacements with reduction. Subjects will have an examination using the CMI at their screening visit. Subjects who meet inclusion criteria will be randomized to one of three groups: The study device (Clayton Intra-aural Device (CID)) group, the mouth splint group, or the exercise group. Subjects in all groups will return to the clinic for a baseline visit, followed by visits at one month, two months and three months post-baseline to return their completed 4 week VAS diary and to complete follow-up testing. At the baseline visit, subjects will have a targeted physical examination, with results documented by the investigator on the CMI questionnaire. Subjects will complete an in-office VAS score, a Modified SSI questionnaire, and will also complete the TMJ Scale, a questionnaire designed to measure possible improvement using a 10 point scale. At each follow-up visit, each subject will complete questionnaires (including the Modified SSI questionnaire and an in-office VAS score)and will have a targeted physical examination, with results documented by the investigator on the CMI questionnaire. At each follow-up visit, subjects will be issued a new monthly diary to complete for the VAS scores twice daily, (once in the morning before 10:00 a.m. and once before bed) as well as to track their device wearing time or exercise compliance, as applicable. At the three month follow-up visit, subjects will also complete the TMJ Scale. Adverse events will be assessed at each visit.

ELIGIBILITY:
Inclusion Criteria:

A subject must meet all of the following criteria to be eligible for study participation:

* Subjects who present to IMIC for jaw pain or dysfunction
* Subjects who sign and date an IRB/EC approved informed consent form
* Subjects must have an RDC/TMD diagnoses that include at least one of the following:

  * Myofascial Pain
  * Arthralgia
  * Disc displacement with reduction; AND

The subject has the presence of one or more of the following findings associated with pain as demonstrated with a VAS score of >4:

* Increased (>60mm) or decreased (<40mm) range of interincisal jaw opening;
* Pain upon any jaw movement;
* Pain on digital palpation (about 0.45 kg of pressure) of the periauricular area or external auditory meatal areas;
* Pain on digital palpation (about 0.45 kg of pressure) in 2 or more muscles of mastication; or
* Joint sound with pain

Exclusion Criteria:

* Subjects diagnosed with rheumatoid arthritis, osteoarthritis, osteoarthrosis or another connective tissue disorder
* Subjects who have had direct trauma to the jaw
* Subjects who have used an occlusal appliance to treat a TMD within the previous six months
* Subjects who have had prior TMJ or ear surgery
* Subjects with any physical or behavioral disorder, which, in the opinion of the Principal Investigator, may interfere with the use of the device or compliance with the study protocol
* Subjects who have a narrow ear canal or impression of the ear canal, which is prolapsed due to an anatomical shift or failure of the ear canal wall structure, or a canal that does not allow for the ear canal second turn to be identified
* Subjects with visible or congenital ear deformity as observed on targeted physical exam
* Subjects whose ear canal anatomy does not allow for fit of the study device
* Subjects who have taken a narcotic pain medication in the last seven days or who have taken aspirin or a non-steroidal anti-inflammatory agent in the last 24 hours
* Subjects who have a history of ear pain unrelated to TMJ
* Subjects who have a history of ear drainage in the past 2 years
* Subjects who have active ear drainage, swelling, or redness as observed on targeted physical exam
* Subjects whom the investigator believes may not be a appropriate candidates for an intra-oral splint due to missing or poor quality dentition or untreated pain of dental origin (pulpal pain, pericoronitis of wisdom teeth, or similar conditions)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2008-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Tsuchiya, DDS, Principal Investigator — Insitituto Mexicano de Investigacion Clinica; Lawrence G. Clayton, M.A., Study Director — Ascentia Health, Inc.
Locations (1):
- Instituto Mexicano de Investigacion Clinica, Mexico City, D.f., Mexico

REFERENCES:
- [Derived] Tavera AT, Montoya MC, Calderon EF, Gorodezky G, Wixtrom RN. Approaching temporomandibular disorders from a new direction: a randomized controlled clinical trial of the TMDes ear system. Cranio. 2012 Jul;30(3):172-82. doi: 10.1179/crn.2012.027. PMID 22916669

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects completed a screening visit and were provided a diary record their Temporomandibular Disorder severity. Subjects returned to the clinic, were randomized if they qualified, and were assigned a treatment group. 150 subjects were planned, but the site over-enrolled 2 subjects due to a temporary problem with the database subject count.
Groups:
- Clayton Intra-aural Device (CID) Group: Treatment group receiving the Clayton Intra-aural Device (CID)
- Mouth Splint Group: Group receiving an intra-oral flat-plane splint
- Jaw Exercise Group: Jaw exercise group, who receive no device but completed a study-specified jaw exercise program
Period: Overall Study
Arm/Group | Clayton Intra-aural Device (CID) Group | Mouth Splint Group | Jaw Exercise Group
Started | 60 | 64 | 28
Completed | 52 | 56 | 22
Not Completed | 8 | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clayton Intra-aural Device (CID) Group | Mouth Splint Group | Jaw Exercise Group | Total
Number analyzed (Participants) | 60 | 64 | 28 | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 60 | 64 | 27 | 151
  >=65 years | 0 | 0 | 1 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 37.29 (10.63) | 38.02 (11.02) | 36.27 (12.97) | 37.41 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 53 | 25 | 126
  Male | 12 | 11 | 3 | 26
Region of Enrollment [Number; unit: participants]
  Mexico | 60 | 64 | 28 | 152

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline In Craniomandibular Index (CMI) Scores At 3 Months (In A Scale)
Description: The Craniomandibular Index (CMI) is designed to provide a basis for evaluating the severity of Temporomandibular Disorder (TMD) signs and symptoms. The assessment involves asking questions related to the condition of Mandibular Movement, TMJ noise, and palpations of the extraoral muscle, neck muscle, TMJ capsule and intraoral muscle. The answers to all of the questions are combined to calculate a score from 0 to 1 in which 0 represents no TMD signs and symptoms and 1 represents the most severe TMD signs and symptoms.
Time Frame: Change from Baseline in Craniomandibular Index (CMI) Scores at 3 months (in a scale)
Population: The arm that includes "0" (Jaw Exercise) is reported in Seconary Outcome Measure Table.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clayton Intra-aural Device (CID) Group | Mouth Splint Group | Jaw Exercise Group
Number analyzed (Participants) | 60 | 64 | 0
Units on a scale | .23 (.21) | .20 (.15) |
Statistical Analysis 1: Comparison: Clayton Intra-aural Device (CID) Group vs Mouth Splint Group; The LS means were used to calculate the test statistic for non-inferiority of the CID to the traditional splint device. The null hypothesis was that the reduction of CMI score for the CID is less than 80% of the reduction in the splint group. A significant p-value(< 0.05) would reject this null hypothesis in favor of the alternative hypothesis that the CID demonstrated a reduction of at least 80% of that seen in the splint group; Test type: Non-Inferiority or Equivalence — The unadjusted reductions are straight arithmetic averages and are supplied for informational purposes only. The pooled variance is calculated from the unadjusted standard deviations, and the t statistic is calculated as described in Laster (2003) using an average sample size of 54 and 106 degrees of freedom; p < 0.0096, student's t-test with 2n-2 DoF

2. Primary Outcome: Number of Subjects With Adverse Events
Description: Subjects were assessed for adverse events from the baseline visit through study completion (3 months post-baseline). Adverse events were categorized by the investigator for severity and relationship to treatment.
Time Frame: From Baseline through 3 months post-baseline visit.
Measure: Number; unit: Participants
Arm/Group | Clayton Intra-aural Device (CID) Group | Mouth Splint Group | Jaw Exercise Group
Number analyzed (Participants) | 60 | 64 | 28
Participants | 11 | 10 | 3
Statistical Analysis 1: Comparison: Clayton Intra-aural Device (CID) Group vs Mouth Splint Group; Safety analyses were performed on the ITT population. The safety of the CID was characterized by the proportion of subjects with all serious and non-serious study-related adverse events and Unanticipated Adverse Device Events (UADEs). In addition, summaries of the onset, duration, severity, treatment relatedness, and outcome of all adverse events were reported; Test type: Non-Inferiority or Equivalence — Safety analyses were performed on the ITT population; p = 0.688, t-test, 1 sided

3. Secondary Outcome: Change From Baseline In Craniomandibular Index (CMI) Scores At 3 Months (In A Scale)
Description: as for outcome 1
Time Frame: Change from Baseline in Craniomandibular Index (CMI) Score at Three Months Post-Baseline (in a scale)
Population: The arm that includes "0" (Mouth Splint Group) is included in the Primary Outcome Measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Clayton Intra-aural Device (CID) Group: This group of subjects received the Clayton Intra-aural Device
- Mouth Splint Group: This group was not part of the analysis
- Jaw Exercise Group: This subject group received no device but was assigned to complete a study-specified jaw exercise program
Arm/Group | Clayton Intra-aural Device (CID) Group | Mouth Splint Group | Jaw Exercise Group
Number analyzed (Participants) | 60 | 0 | 28
Units on a scale | .23 (.21) |  | .15 (.13)
Statistical Analysis 1: Comparison: Clayton Intra-aural Device (CID) Group vs Jaw Exercise Group; A significant p-value for the treatment group effect would indicate that the CID group and Exercise group were significantly different, based on results of a two-sided t test for difference in means, with alpha=0.5, and allowing for unequal sample sizes; Test type: Superiority or Other; p = .2995, t-test, 2 sided — From the pilot study, 50 subjects (CID arm) and 25 (exercise arm) were required for at least 80% power to detect a difference in the mean reduction in CMI scores between arms if muPassive is less than approximately 70% of that in the CID arm

ADVERSE EVENTS:
Time Frame: Continuous, from baseline through study exit.
Description: After consent, the baseline visit was the point at which adverse event reporting began. Adverse events were collected continuously throughout the study until individual subject study exit.
Arm/Group | Clayton Intra-aural Device (CID) Group | Mouth Splint Group | Jaw Exercise Group
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/64 | 0/28
Other Adverse Events (participants affected / at risk) | 7/60 | 9/64 | 3/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clayton Intra-aural Device (CID) Group (N=60) | Mouth Splint Group (N=64) | Jaw Exercise Group (N=28)
Discomfort or Pain (General disorders) | 4 (5) | 6 (7) | 2 (2)
Headache (General disorders) | 3 (3) | 3 (6) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No